CLINICAL TRIAL: NCT07314567
Title: An Open Label, Single Arm Study to Assess Safety, Efficacy and Persistence of ACE1831, in Subjects With Relapsed/Refractory Systemic Lupus Erythematosus (SLE)
Brief Title: ACE1831 in Adult Subjects With Relapsed/Refractory Systemic Lupus Erythematosus （SLE）
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lingli Dong, Director of the department of rheumatology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE1831-301
Record Dates: First submitted 2025-11-26; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: System Lupus Erythematosus(SLE)
Keywords: ACE1831; SLE; Refractory Systemic lupus erythematosus (SLE); gamma delta T (gdT) cell
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant (Experimental): The single, open label study arm includes 2 dose escalation cohorts:
  Cohort 1: Receives ACE1831 (Dose Level 1) with LDC depending on assignment Cohort 2: Receives ACE1831 (Dose Level 2) with LDC depending on assignment
  Interventions: Drug: ACE1831; Drug: Lymphodepleting chemotherapy

INTERVENTIONS:
Drug: ACE1831 — ACE1831 is allogeneic gamma delta T (gdT) cell therapy. Subjects will receive ACE1831 dose based on the assigned dose escalation cohort.
Drug: Lymphodepleting chemotherapy — Subjects assigned to receive lymphodepleting preconditioning (LDC) will receive chemotherapy cyclophosphamide ahead of ACE1831 administration.

SUMMARY:
ACE1831 is an off-the-shelf, allogeneic gamma delta T (gdT) cell therapy derived from healthy donors, that is under investigation for the treatment in subjects with Relapsed/Refractory Systemic lupus erythematosus (SLE)

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 60 years (inclusive)
* History of meeting the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria, or the 1997 ACR criteria, or the 2012 Systemic Lupus International Collaborating Clinics (SLICC)
* Presence of anti-dsDNA antibodies and/or anti-nuclear antibodies (ANA) and/or anti-Smith (anti-Sm) antibodies positive
* SLE is in the moderate to severe active phase with the SLEDAI-2000 score ≥ 8
* At least one British Isle Lupus Rating Group Index (BILAG-2004) Class A (severe manifestation) or two Class B (moderate manifestation) organ scores, or both
* Inadequate response to glucocorticoids and at least 2 of treatments used for at least 3 months
* Women of childbearing potential and their partners must agree to use at least 1 highly effective method of contraception throughout the study period and for 1 year after treatment
* Signed informed consent

Exclusion Criteria:

* Severe lupus nephritis requiring prohibited medications for active nephritis treatment，or hemodialysis, or eGFR < 50 ml/min/1.73m²
* Central nervous system disease caused by SLE or other conditions
* Significant medical history that would pose a risk to the patients safety from the investigator's opinion, or patients medical condition could worsen during the study
* Malignancies within 5 years
* Presence of active, recurrent, chronic infection requiring treatment , or latent infection (HBV, HCV, HIV, TB, syphilis)
* Received any B-cell depletion biologic therapy
* Received immunosuppressive small molecule drug therapy， or other systemic corticosteroid therapy ， or prednisone
* Pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ACE1831 in subjects with Refractory Systemic lupus erythematosus | 24 weeks after last dose of ACE1831
  To assess the incidence of Adverse Events (AEs), [AEs including Treatment Emergent AEs, Serious AEs (SAEs), AEs of Special Interests (AESIs), and dose limiting toxicities (DLTs)] (unit: number of AEs)

SECONDARY OUTCOMES:
To assess the efficacy of ACE1831： Changes in SLE disease activity Index (SLEDAI-2000) score | 24 weeks after last dose of ACE1831
  Changes of SLE disease activity Index (SLEDAI-2000) score
To assess the efficacy of ACE1831 (secondary efficacy)：Changes in PGA | 24 weeks after last dose of ACE1831
  Changes in Physician's Global Assessment (PGA) of disease activity score (Visual Activity Score,scale range 0 - 100)
To assess the efficacy of ACE1831 : Changes in SGA | Time Frame: 24 weeks after last dose of ACE1831
  Changes in Subject's Global Assessment (SGA) of disease activity score (Visual Activity Score,scale range 0 - 100)
To assess the efficacy of ACE1831 ：Changes in LupusQOL | 24 weeks after last dose of ACE1831
  Changes of Lupus Qualituy of Life(LupusQOL) total score
To assess the efficacy of ACE1831 ：Changes in EQ-5D-5L score | 24 weeks after last dose of ACE1831
  Changes of European Quality of Life Five Dimension Five Level questionnaire(EQ-5D-5L )score
To assess the efficacy of ACE1831 ：Changes in SF-12 score | 24 weeks after last dose of ACE1831
  Changes in Quality of Life Questionnaire (QOL) Short Form 12 (SF-12) total score
To assess the efficacy of ACE1831 ：Changes in BILAG-2004 score | 24 weeks after last dose of ACE1831
  Changes of BILAG-2004 score
To assess the efficacy of ACE1831: LLDAS rate | 24 weeks after last dose of ACE1831
  Proportions of subjects achieving LLDAS by timepoint
To assess the efficacy of ACE1831: DORIS | 24 weeks after last dose of ACE1831
  Proportions of subjects who achieved remission according to the DORIS by timepoint
To assess the efficacy of ACE1831: SRI-4 response rate | 24 weeks after last dose of ACE1831
  Proportion of participants who achieved Systemic Lupus Erythematosus Responder Index -4 (SRI-4) response
Persistence of ACE1831 after administration | 8 weeks after last dose of ACE1831
  Half-life of ACE1831
Measure the pharmacodynamics change of ACE1831 | 24 weeks after last dose of ACE1831
  Immunoglobulin, cytokines, lymphocytecount , autoantibody titers, complement C3 and C4 levels, C-reactive protein, erythrocyte sedimentation rate, etc
Immunogenicity | 24 weeks after last dose of ACE1831
  Titration of anti-ACE1831 antibodies after administration

OTHER OUTCOMES:
To assess the efficacy of ACE1831： single-cell sequencing | 24 weeks after last dose of ACE1831

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No